CLINICAL TRIAL: NCT07160543
Title: Non-Immersive Virtual Environments for the Treatment of Hoarding Disorder: A Preliminary Randomized Controlled Trial With a Mixed Factorial Design Based on a Non-Clinical Sample
Brief Title: Non-Immersive Virtual Environments for the Treatment of Hoarding Disorder
Acronym: HD&VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DD0A28FFB2B4C63CFED6CC9BACC7A5
Record Dates: First submitted 2025-08-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-05

CONDITIONS: Hoarding Disorder; Virtual Reality Based Therapy; General Population (no Specific Condition or Disease)
MeSH Terms: conditions — Hoarding Disorder; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: participants were randomly assigned to one of the two experimental conditions. Randomization was conducted using a simple, computer-generated sequence via the "RAND" function in Excel, ensuring allocation concealment. The randomization was unrestricted, meaning no blocking or stratification procedures were employed. This approach ensured that each participant had an equal probability of assignment to either condition, regardless of enrollment order or participant characteristics. The random allocation sequence generation and participant enrollment were performed by two master 's-level psychology students. Blinding procedures were implemented to reduce bias. Although participants were aware of the intervention they received due to the nature of the exposure tasks, outcome assessors were blinded to group allocation. The researchers responsible for data analysis and interpretation were not involved in the delivery of the interventions and did not have access to identifying participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Imagination Exposure Condition (Active Comparator): Participants were asked to close their eyes and vividly imagine discarding the personal object they had previously selected. The procedure was guided verbally by the experimenter, who instructed participants to mentally visualize moving the object from their personal space to a trash bin. The aim was to evoke the emotions and cognitive reactions associated with discarding in a controlled, internalized format. Intervention Assigned: Behavioral: Imagination Exposure.
  Interventions: Behavioral: Imagination Exposure
- Arm 2: Non-immersive Virtual Reality Exposure Condition (Experimental): Participants interacted with a non-immersive, computer-based virtual environment displayed on a standard monitor. The environment simulated a household setting with various rooms and a trash bin located in a virtual garage. Participants navigated the space using a keyboard and mouse. They were presented with a digital representation of their own personal object, which had been previously photographed and embedded into the virtual scene. They were instructed to drag the object into the virtual trash bin, simulating the act of discarding. Intervention Assigned: Device: Non-immersive Virtual Reality Exposure.
  Interventions: Device: Non-immersive Virtual Reality Exposure

INTERVENTIONS:
Behavioral: Imagination Exposure — Participants were guided to close their eyes and imagine discarding their personal object. The experimenter provided standardized verbal instructions to help participants visualize moving the item from their own space into a trash bin.
  Other Names: IE; Imagination-based Exposure
  Arms: Arm 1: Imagination Exposure Condition
Device: Non-immersive Virtual Reality Exposure — Participants used a desktop computer to interact with a virtual household environment. Their personal object, photographed beforehand, was digitally embedded in the scene. Using keyboard and mouse, participants navigated to the virtual garage and dragged the object into a virtual trash bin. The experimenter remained present to provide support.
  Other Names: VRE; Virtual Reality Exposure; Computer-based VR
  Arms: Arm 2: Non-immersive Virtual Reality Exposure Condition

SUMMARY:
This experimental trial investigates whether Virtual Reality Exposure (VRe) helps individuals reduce the difficulty of discarding personal possessions. It will also evaluate the psychological state impacts of the intervention. The main questions it aims to answer are:

Does exposure-based intervention (VRe) reduce emotional distress and improve willingness to discard personal items? What psychological reactions (such as anxiety or emotional responses) do participants experience during and after these interventions?

DETAILED DESCRIPTION:
Researchers will compare the effects of VRe to Imagination exposure (Ie) to determine which method is more effective in reducing discarding-related difficulties. The trial is specifically designed for individuals from the general population who do not meet the criteria for hoarding disorder but experience significant emotional discomfort when trying to part with certain belongings. This subclinical presentation of hoarding-like behavior is common and often unaddressed despite its impact on well-being and living space management.

Participants completed online assessments and screening procedures to determine eligibility. They then participated in a one-time, in-lab exposure session using VRe or Ie techniques. Based on a standardized rating scale, each participant brought a personal object they had previously identified as difficult to discard but not overly emotionally charged. During the session, they engaged in either an immersive visualization of discarding the item (Ie) or a guided interaction with a virtual simulation of discarding the item (VRe). Participants were evaluated on psychological (e.g., state anxiety, positive and negative affect) and behavioral outcomes (e.g., actual discarding behavior) before and after the exposure. At the end of the session, participants reported whether they intended to discard the physical object in real life.

This study follows a single-session randomized controlled trial (RCT) design with partial blinding of outcome assessors. While participants were aware of the intervention type they received due to the nature of the exposure task, the researchers responsible for scoring and analyzing outcome data were blinded to group allocation to minimize bias and expectancy effects. This design enhances the rigor and objectivity of outcome comparisons between groups.

This preliminary RCT adopts an exploratory approach due to the limited empirical research on using non-immersive VR for discarding behaviors, particularly in non-clinical populations. Prior findings suggest that VR-based interventions can simulate real-world behavior and reduce emotional reactivity in anxiety-related contexts. However, existing studies have primarily focused on immersive VR applications and clinical populations, such as individuals with specific phobias or PTSD. The current study aims to fill this gap by assessing the potential of non-immersive, more accessible VR platforms in promoting behavioral change related to possession management.

The specific objectives of the study are:

To investigate whether exposure to a non-immersive VR environment can help individuals discard personally relevant objects more effectively than imagination-based exposure; To assess within- and between-group differences in emotional and behavioral responses-specifically state anxiety, positive and negative affect, and discarding behavior-before and after the intervention.

Given the preliminary nature of this research, the following two hypotheses guide the investigation:

Hypothesis 1: Participants in the VR exposure condition will be more likely to discard their object during or after the session than participants in the imagination-based exposure group. This hypothesis is grounded in preliminary evidence suggesting that non-immersive VR can support emotional regulation and task engagement by providing a structured yet low-pressure simulation of real-world scenarios.

Hypothesis 2: Both groups will show a reduction in state anxiety and negative affect, along with a potential increase in positive affect, from pre- to post-exposure. However, participants in the VR condition may exhibit greater improvements due to the virtual environment's interactive and visually grounded features, which may facilitate emotional processing and cognitive restructuring.

ELIGIBILITY:
Inclusion Criteria:

Adults individuals from general population.

Exclusion Criteria:

* A score of 4 or higher on the self-report item of the Hoarding Rating Scale Self-Report, which assesses difficulty in discarding possessions;
* No evident signs of suicidal ideation, based on the scores of the Beck Depression Inventory-II, nor indications of alcohol or substance abuse, psychotic spectrum disorders, depressive disorders, organic mental disorders, or conditions associated with cognitive impairment;
* Participants must report difficulty in discarding certain objects. Moreover, individuals have to complete online monitoring questionnaires via PC or smartphone.
* Participants had to fill out a custom questionnaire evaluating each object based on two parameters: importance and difficulty in discarding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in State Anxiety as measured by the State-Trait Anxiety Inventory (Y)- State subscale | Baseline (immediately before the intervention) and Post-intervention (immediately after completion of the single experimental session).
  State anxiety is a psychological feature focused on how individuals experience at particular times (state anxiety). It will be assessed using the State subscale of the "State-Trait Anxiety Inventory (STAI-Y) State subscale", a validated self-report questionnaire commonly used in clinical and experimental research to measure transient levels of anxiety. Scores range from 20 to 80, with higher scores indicating greater state anxiety.
Change in Positive and Negative Affect as measured by the Positive and Negative Affect Schedule (PANAS) | Baseline (immediately before the intervention) and Post-intervention (immediately after completion of the single experimental session).
  Positive and negative affect will be assessed using the Positive and Negative Affect Schedule (PANAS), a validated self-report questionnaire consisting of 20 items. The scale includes two subscales: Positive Affect (10 items; scores range 10-50) and Negative Affect (10 items; scores range 10-50). Higher scores indicate greater intensity of the corresponding affective state.
Frequency of Discarding Behavior (Behavioral Observation) | During the single experimental session (immediately after intervention).
  Discarding behavior was assessed through direct behavioral observation during the experimental task. The measure consisted of recording whether participants discarded the personal object (in the imagination condition or in the virtual reality condition) and the frequency of this behavior within the single session.

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Novara, PhD, Principal Investigator — University of Padova; Susanna Pardini, PhD, Principal Investigator — Centre for Digital Health and Well-being, Fondazione Bruno Kessler, Trento, Italy
Locations (1):
- University of Padova, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No